CLINICAL TRIAL: NCT02961933
Title: Utah Study Evaluating Apneic Oxygenation for Emergency Department Intubation
Acronym: USE AP OX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1050200
Record Dates: First submitted 2016-11-01; First posted 2016-11-11 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Intubation
Keywords: hypoxemia; intubation; apneic oxygenation
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apneic oxygenation (Experimental)
  Interventions: Other: Apneic oxygenation
- non-apneic oxygenation (Active Comparator)
  Interventions: Other: Pre-oxgenation with NRB, NIPPV, BVM

INTERVENTIONS:
Other: Apneic oxygenation — Nasal cannula apneic oxygenation
  Arms: Apneic oxygenation
Other: Pre-oxgenation with NRB, NIPPV, BVM — Pre-oxygenation with non-rebreather mask, non-invasive positive pressure ventilation, or bag-valve mask
  Arms: non-apneic oxygenation

SUMMARY:
This study will determine rates of first pass success without hypoxemia in emergency department intubations with and without the use of apneic oxygenation by nasal cannula.

ELIGIBILITY:
Inclusion Criteria:

- Patients requiring emergent Rapid Sequence or Delayed Sequence endotracheal intubation with administration of a neuromuscular blocker (Succinylcholine, Rocuronium)

Exclusion Criteria:

* Known prisoners
* Patients in cardiac arrest
* Patients who are intubated without the use of neuromuscular blockade (i.e., cardiac arrest, awake intubation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2016-12; Primary Completion 2020-01 (Actual); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
First pass success without hypoxemia | 10 minutes

SECONDARY OUTCOMES:
Change in peri-intubation saturation | 0, 30, 60 and 120 seconds
Saturation at time of tube placement | 10 minutes
Time to desaturation <93% | measured time until saturations drop below 93% during the peri-intubation period, up to 10 minutes
Saturation at post intubation | 0, 30, 60, and 120 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bryant, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No